CLINICAL TRIAL: NCT04123574
Title: A Pilot Proof of Mechanism Study of BXCL701, a Small Molecule Inhibitor of Dipeptidyl Peptidases (DPPs), in Patients With Pancreatic Cancer
Brief Title: A Pilot Study of BXCL701 in Patients With Pancreatic Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No longer relevant to field
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXCL701-001
Record Dates: First submitted 2019-04-30; First posted 2019-10-11 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cancer of Pancreas; Cancer of the Pancreas; Neoplasms, Pancreatic; Pancreas Cancer; Pancreatic Cancer
Keywords: Pancreas; Cancer; Neoplasms; Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — PT-100 dipeptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): BXCL701 will be administered for one week at a dose of 0.2 mg, twice daily (BID). If BXCL701 is well-tolerated after the first week of treatment, the dose will be increased to 0.3mg BID for a total daily dose of 0.6mg to all patients for the second week of treatment.
  Interventions: Drug: Talabostat Mesylate

INTERVENTIONS:
Drug: Talabostat Mesylate — BXCL701 tablets dosage strengths include 0.2mg and 0.05mg tablets for oral administration.
  Patients are to self-administer the prescribed number of BXCL701 tablets for a total daily dose of 0.6 mg. BXCL701 should not be taken on an empty stomach.
  Daily blood pressure monitoring will be performed during the dosing period. Administration of at least 1L of intravenous (IV) fluids is required on Day 1.
  On days when pharmacokinetic (PK) assessments are being performed, BXCL701 should be administered at the study center and should be administered at (approximately) the same time of day on each treatment day.
  Other Names: BXCL701

SUMMARY:
A study to assess the biochemical and immunomodulatory effects of BXCL701 in pancreatic cancer.

DETAILED DESCRIPTION:
This is a Phase 0 or "window of opportunity" study where paired specimen analysis, taken before and after drug exposure, will permit the evaluation of target modulation and assessment of immune effector cell infiltration into the tumor and the generation of relevant immune cytokines.

In this study, BXCL701 will be administered at a dose of 0.3 mg, twice daily for a total daily dose of 0.6mg (the previously defined maximum tolerated dose [MTD] of the drug), to all patients for a short period of 14 days. This study is designed to assess the biochemical and immunomodulatory effects of BXCL701 in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Has untreated (eg, no prior investigational therapies, chemotherapy, or radiation therapy), locally advanced or metastatic adenocarcinoma of the head, neck, uncinate process, or tail of the pancreas with a local or metastatic lesion that is amenable to biopsy before and after treatment. (Whenever possible, the before and after treatment biopsies should be from the same lesion.)
2. Is able and willing to undergo tumor biopsy before and after treatment. (A pretreatment biopsy may not be needed if tissue is available from a biopsy conducted within 28 days prior to screening that is adequate for the study assessments.)
3. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Is 18 to 75 years of age, inclusive
5. Has adequate organ function within 28 days of treatment initiation
6. For participants with exposure to prior agents associated with decreased left ventricular ejection fraction (LVEF) (e.g. anthracyclines), or if clinically warranted, a documented LVEF > 45% using a standard echocardiogram (ECHO) or multigated acquisition (MUGA) scan test at Screening or within 60 days prior to Cycle 1 Day 1. ECHO or MUGA testing for other participants without relevant medical history or clinical symptoms can be performed if feasible.
7. Has oxygen saturation ≥ 92% on room air.
8. Is able to take an oral medication.
9. Has signed an Informed Consent Form (ICF) prior to the initiation of any study-specific procedures or treatment.
10. Is willing and able to adhere to the study visit schedule and other protocol requirements.
11. Women of childbearing potential (WOCBP) must have a negative pregnancy test at baseline. A woman must be menopausal for at least 12 months before she is considered not to be of reproductive potential.
12. Male and female patients of reproductive potential must agree to use an effective contraceptive method during participation in this study and for 6 months following the study.

Exclusion Criteria:

1. A female who is pregnant or breast-feeding.
2. Has other concurrent malignancies except for basal and squamous cell cancers of the skin and in-situ cervical cancer.
3. Has uncontrolled epilepsy, central nervous system diseases, or a history of mental disorder that is severe enough to hinder the ability of the patient to provide informed consent or that may influence the patient's compliance with the protocol in the judgments of the investigator.
4. Has an upper gastrointestinal obstruction, abnormal physiological function, or malabsorption syndrome that may affect the absorption of study medication.
5. Has required chronic corticosteroids, defined as > 10 mg/day of prednisone or equivalent, or immunosuppressive therapy within the past 3 months. Patient requires treatment with DPP4 inhibitors (e.g. gliptins).
6. Has a premalignant hematologic disorder, eg, myelodysplastic syndrome.
7. Has a severe organ dysfunction or disease that might prevent completion of the treatment regimen, eg, cardiopulmonary diseases (New York Heart Association [NYHA] ≥ Class III, arrhythmia Lown III/IV, global respiratory insufficiency); ascites; acute pancreatitis; bleeding diathesis, coagulopathy, or need for full dose anticoagulation.
8. Has a chronic infectious disease, especially immune deficiency syndromes, eg, human immunodeficiency virus (HIV) infection, active tuberculosis within 12 months prior to potential study participation or suspected/active SARS-CoV-2 (Covid-19) infection.
9. Has a history of severe neurologic disorders, eg, cerebrovascular ischemia within the past year.
10. Has a history of prior deep venous thrombosis or pulmonary embolism within the past year.
11. Has serious medical, psychological, familial, sociological, or geographical conditions or circumstances potentially hampering compliance with the study protocol and follow-up.
12. QT interval corrected for heart rate using Bazett's formula (QTcB) > 440 msec at Screening.
13. Patients with history of symptomatic orthostatic hypotension within 3 months prior to enrollment. Orthostatic hypotension is defined as a drop in systolic blood pressure (BP) of ≥ 20 mmHg or diastolic BP of ≥ 10 mmHg with assumption of an upright posture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2021-12-06 (Estimated); Study Completion 2021-12-06 (Estimated)

PRIMARY OUTCOMES:
To characterize the quantitative and qualitative effects of BXCL701 on relevant immune effector cytokines and various immunological effector cells that are consistent with its known mechanism of action. | Up to 37 days post treatment
  To measure how BXCL701 effects the tumor by measuring the rate of tumor cell death or the reduction of tumor cell growth. This will be measured by scans and blood work.

SECONDARY OUTCOMES:
Evaluate the tolerability of exposure to BXCL701: National Cancer Institute Common Terminology Criteria | Up to 37 days post treatment
  assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events
Evaluate the effect of exposure to BCXL701 on cancer cell death | Up to 37days post treatment
  Measure the rate of cancer cell death measured by histological staining methods of post-treatment biopsied tissue.
Genomic analysis before and after treatment. | Up to 37 days post treatment
  Genomic analysis is the identification, measurement or comparison of genomic features such as DNA sequence, structural variation, gene expression, or regulatory and functional element annotation at a genomic scale.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - BioXcel Clinical Research Site, Boston, Massachusetts
  - BioXcel Clinical Research Site, New York, New York

IPD SHARING:
Plan to Share IPD: No